CLINICAL TRIAL: NCT06651372
Title: Interest of Systematic Screening for Dengue, Chikungunya, and Zika, in Patients for Whom a Malaria Diagnosis is Negative, in the Event of a Recent Return From Travel: a Retrospective Study at the University Hospitals of Strasbourg, 2024-2025
Brief Title: The Interest of Systematic Screening for Dengue, Chikungunya, and Zika, in Malaria-negative Return Travelers
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: IV-0198
Record Dates: First submitted 2024-10-17; First posted 2024-10-21 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Arbovirus Infections
Keywords: Post-travel infections; Dengue; Chikungunya; Zika disease; Arbovirus screening
MeSH Terms: conditions — Arbovirus Infections; Dengue; Chikungunya Fever | interventions — Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Malaria negative return travelers: Any person, man or woman, aged over 18, treated at the University Hospitals of Strasbourg from January 2024 to December 2025, having received a blood sample as part of the treatment, for a diagnosis of malaria upon return from a recent trip whose result was negative. Any person who has already consented or has not objected to their biological resources being preserved in the "Microbiology" biocollection and reused for scientific research.
  Interventions: Biological: The retrospective analyses planned for these samples consist of serological analysis and molecular analysis (RT-PCR ) according to the date of symptoms ons

INTERVENTIONS:
Biological: The retrospective analyses planned for these samples consist of serological analysis and molecular analysis (RT-PCR ) according to the date of symptoms ons — Serological tests detecting IgM and IgG

SUMMARY:
International travel has increased dramatically in recent years. Vector-borne pathologies such as malaria and arboviruses are common etiologies of post-travel fever, which are prevalent in similar geographical areas (tropical and intertropical). Arboviruses, for "arthropod-borne viruses," are transmitted by the bite of blood-sucking vectors (mosquitoes, ticks, or sandflies). The dengue, chikungunya, and zika viruses are transmitted through the bite of an infected Aedes mosquito (Aedes aegypti and Aedes albopictus).

The establishment of Aedes albopictus (tiger mosquito), competent for transmitting these 3 viruses, since 2004 in mainland France and the transit of travelers carrying a virus allowed the appearance of the first autochthonous cases of dengue and zika. Each year, outbreaks of autochthonous cases of dengue fever are reported in the PACA, Occitanie, and Auvergne-Rhône Alpes regions, and a cluster of 3 Indigenous cases was reported in 2023 in the Paris region.

Since 2014, the tiger mosquito has been established in Bas-Rhin. Between 2014 and 2022, the vector was detected in around thirty municipalities around Strasbourg. In a department where the spread of the tiger mosquito is evolving rapidly, these data remind us that only an early diagnosis, delivered quickly, allows effective vector control measures to avoid generating autochthonous transmission.

In a previous study carried out at the Virology laboratory, we retrospectively analyzed the diagnosis of these 3 arboviruses after the exclusion of malaria in the context of recent travel over a period of 10 years (2014-2023). Among the 913 patients included, for 78% of cases (n=714), no testing for dengue, chikungunya, or zika was carried out, a proportion stable over 10 years.

These three arboviruses seem underdiagnosed, and we assume, given our previous results, that 8 to 10% of patients for whom, in the context of recent travel, a test for malaria comes back negative are imported cases of dengue, chikungunya, or zika. At the end of this retrospective study, we want to evaluate this sub-diagnosis on a larger sample to propose a review of practices and the establishment of Arbovirus-malaria "reflex testing." Currently, no French or similar European data is available, allowing us to evaluate this under-diagnosis, which constitutes a significant risk of the emergence of indigenous clusters in our territory.

The main objective of this study is to determine the infection rate by dengue, chikungunya, and zika viruses identified when the diagnosis is made after the exclusion of negative malaria in the context of recent travel among patients treated at the Strasbourg University Hospitals between January 1, 2024, and December 31, 2025.

The secondary objectives of this work are as follows:

Estimate the prevalence of different clinical symptoms (patient medical records) in retrospectively identified cases of dengue, chikungunya, and zika.

* Evaluate the onset time of symptoms in relation to the date of return/arrival from the area of stay of retrospectively identified cases of dengue, chikungunya, and zika.
* Evaluate the delay in the appearance of symptoms in relation to the date of taking the initial sample (the one leading to the diagnosis of negative malaria) of retrospectively identified cases of dengue, chikungunya, and zika.
* Study the laboratory results associated with the initial management of the patient (biochemical assessment and blood count) of retrospectively identified cases of dengue, chikungunya, and zika.
* Study the distribution of areas, periods, and reasons for staying in retrospectively identified dengue, chikungunya, and zika cases.

Study the municipalities of residence of positive cases in the areas where the tiger mosquito is established.

ELIGIBILITY:
Inclusion criteria:

* Adult subject (≥18 years old), man or woman
* Supported at Strasbourg University Hospital between 01/01/2024 and 12/31/2025
* Having received a blood sample as part of the treatment for which the test for malaria was negative, following a recent return from a trip (≤ 31 days)
* Having already given their consent for their biological resources to be preserved in the "Microbiology" biocollection and reused for scientific research purposes.

Exclusion criteria:

* Minor subject (< 18 years old)
* Adult patient for whom a test for malaria came back positive during initial treatment
* Patient having expressed his opposition to participating in the study
* Inability to provide the subject with informed information (subject in an emergency situation, difficulty understanding the subject, etc.)
* Subject under judicial protection
* Subject under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any person, man or woman, aged over 18, treated at the University Hospitals of Strasbourg from January 2024 to December 2025, having received a blood sample as part of the treatment, for a diagnosis of malaria upon return from a recent trip whose result was negative. Any person who has already consented or has not objected to their biological resources being preserved in the "Microbiology" biocollection and reused for scientific research.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
The detection rate of dengue virus, zika virus, or chikungunya virus infection in samples from the subjects studied. | 36 months
  Patients and samples will be selected based on diagnostic activity data from the Medical Mycology Parasitology laboratory. The corresponding production statistics will be produced using the laboratory information system (LIS), glims software from 01/01/2024 to 12/31/2025.
  The retrospective analyses planned for these samples will all be carried out within the microbiology technical platform by the Virology laboratory without any sample transfer.
  Serological tests detecting IgM and IgG will be carried out using the following commercial ELISA kits:
  * Vidas® Anti-chikungunya IgM and IgG
  * Vidas® Anti-dengue IgM and IgG
  * Virclia® Anti-Zika IgM and IgG NS1 antigen detection will be carried out using the Abbott® Bioline Dengue duo test.
  RT-PCR will be carried out using the following kits: EVAg Primers, Probes (Lyoph-P&P) and Positive control for dengue virus detection, chikungunya virus detection and zika virus detection (adapted to Hologic PantherFusion OpenAccess).

SECONDARY OUTCOMES:
Distribution of the clinical symptoms and the biological findings | 36 months
  To estimate the prevalence of different clinical symptoms (patient medical records) in retrospectively identified cases of dengue, chikungunya and zika.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg - Laboratoire de Virologie, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided